CLINICAL TRIAL: NCT05817695
Title: Effect of Different Pacing Sites on Cardiac Synchronization and Tricuspid Regurgitation After Leadless Pacemaker Implantation
Brief Title: Cardiac Synchronization and Tricuspid Regurgitation With Leadless Pacemaker
Acronym: MICRA-SYNK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: MICRA-SYNK-001
Record Dates: First submitted 2023-02-16; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-12

CONDITIONS: Bradycardia
Keywords: Leadless pacing; Synchronization
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Leadless pacemaker — To observe the effect of pacemaker implantation at different sites on cardiac synchronization and tricuspid regurgitation

SUMMARY:
Comparison of cardiac synchronization and tricuspid regurgitation with or without leadless pacemaker pacing in different site

DETAILED DESCRIPTION:
Right ventricular pacing might lead to pacing-induced cardiomyopathy by dyssynchrony and tricuspid regurgitation. Pacing at various sites had different effects on synchrony and tricuspid regurgitation. This study is to observe the effect of leadless pacemaker implantation in different regions on ventricular synchronization and tricuspid regurgitation. Ultrasound and ECG parameter indices are applied.

ELIGIBILITY:
Inclusion Criteria:

patients consent to LP implantation surgery

Exclusion Criteria:

1. Patients with inferior vena cava thrombus, a cancer thrombus, an abnormal inferior vena cava;
2. Patients with femoral vein stenosis and tortuosity failed to accommodate the pacemaker delivery system;
3. Patients with myocardial infarction;
4. Patients who have been implanted with devices that affect the pacemaker delivery system, such as vena cava filters or tricuspid valve mechanical valves;
5. cannot understand or are unwilling to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients consent to LP implantation surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
The evaluation of cardiac electrical synchrony | 1 month
  the QRS duration after pacing
The evaluation of cardiac mechanical synchrony | 1 month
  ①Synchronization analysis between left and right ventricles: interventricular mechanical delay (IVMD) in millisecond.
  ②Left ventricle synchrony analysis: septal-to-posterior wall motion delay (SPWMD) in millisecond，left pre-ejection interval(LPEI) in millisecond.

SECONDARY OUTCOMES:
Age may affect synchronization | 1 month
  Age in years
BMI may affect synchronization | 1 month
  BMI in kg/m^2
Blood pressure may affect synchronization | 1 month
  Systolic and diastolic blood pressure in mmHg
The pacemaker sensing may affect synchronization | 1 month
  pacemaker sensing in millivolt
The pacemaker lead impedance may affect synchronization | 1 month
  lead impedance in ohm

CONTACTS AND LOCATIONS:
Overall Officials: Yi zhou XU, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Yi zhou XU, Hangzhou, Zhejiang, China